CLINICAL TRIAL: NCT06374706
Title: Effects of End-Effector Type Rehabilitation Robots-Morning Walk on Symmetrical Walking Patterns in Individuals With Hemiparesis
Brief Title: Effects of Rehabilitation Robots-Morning Walk in Individuals With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0129
Record Dates: First submitted 2024-03-24; First posted 2024-04-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Healthy Volunteers
Keywords: End-Effector Robot-Morning Walk; Constrained Induced Movement Therapy; Hemiparesis; Symmetry
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Walk Training for Stroke (Experimental)
  Interventions: Behavioral: Morning Walk training for stroke
- Morning Walk Training for Healthy (Active Comparator)
  Interventions: Behavioral: Morning Walk training for healthy

INTERVENTIONS:
Behavioral: Morning Walk training for stroke — Assessing the Feasibility of the End-Effector Rehabilitation Robot, Morning Walk Training and investigate the Immediate Post-Adaptation Effect of Morning Walk Training for Symmetrical Walking on the Ground.
  Arms: Morning Walk Training for Stroke
Behavioral: Morning Walk training for healthy — Assessing the Feasibility of the End-Effector Rehabilitation Robot, Morning Walk Training and investigate the Immediate Post-Adaptation Effect of Morning Walk Training for Asymmetrical Walking on the Ground.
  Arms: Morning Walk Training for Healthy

SUMMARY:
In this study, our objective is to explore and evaluate interventions to improve the process of recovery following a stroke. The main focus is on enhancing symmetrical walking patterns in adults who have experienced neurological deficits due to a stroke. The primary tool will be an end-effector type rehabilitation robot, the Morning Walk®. This robot has been specifically designed to assist in enhancing symmetrical walking patterns for individuals recovering from a stroke Morning Walk® has received approval from the FDA, meaning it meets stringent safety and efficacy standards.

DETAILED DESCRIPTION:
Total forty participants (20 stroke vs 20 healthy individuals) will sign a consent form that is pre-approved by the Institutional Review Board at the participating facilities, which states the purpose of the study, an explanation of the procedures, benefits and risks for the participant, a confidentiality statement, and a refusal/withdrawal policy.

This study will assess the feasibility of end-effector rehabilitation robots, specifically Morning Walk®, to optimize training outcomes and improve symmetry in individuals with stroke.

1. Access the severity of functional and balance capacity prior to gait training. Stroke or healthy participants will first be asked questions about their medical history, physical functionality, and overall well-being. Participants will be equipped with an armband or chest strap to monitor their heart rate. Functional capacity will be assessed using walking tests on the Zeno Walkway system, which evaluates gait speed and spatiotemporal gait parameters during overground walking trials. During the testing process, participants will be recorded on video.
2. Develop the training protocol for the end-effector rehabilitation robot, Morning Walk.

   Prior to the end-effector robot training, Investigators will attach six Delsys wireless electromyographic sensors (Delsys Inc, Natick, MA) to analyze muscle activity in the lower extremities. Additionally, stroke or healthy participants will be equipped with the Tekscan In-Shoes system (Tekscan, Inc., South Boston) to assess temporal events related to foot positioning during training, such as limb loading time. During the end-effector robot training, a saddle-type weight support and secure strap system will be employed to prevent loss of balance or falls. Following an appropriate warm-up and familiarization with the end-effector robot training, various walking parameters of Morning Walk, such as pace, stride length, step height, and initial contact angle, will be examined to achieve balanced loading times between the paretic and non-paretic sides in stroke participants. Training parameters such as step length, step height, and joint angle can be independently adjusted for the paretic and non-paretic sides in stroke patients, and for the dominant and non-dominant sides in healthy individuals. This approach allows for the restriction of movement in the non-paretic or non-dominant side, thereby encouraging the activity of the paretic or dominant side during training. The adaptation training parameters will be adjusted according to the participant's walking capacity. During the training session, participants will be recorded on video.
3. Assessing the Immediate Post-Adaptation Effect of Morning Walk Training on the Ground.

Stroke or healthy participants will be asked to on the Zeno Walkway system to evaluate gait speed and spatiotemporal gait parameters during overground walking trials. During the testing process, participants will be recorded on video.

ELIGIBILITY:
Inclusion Criteria:

* For this study, twenty volunteers fulfilling the inclusion criteria from participating physical therapy facilities and the local community will be recruited. The criteria for participants with a history of stroke include: Age 20 or older.
* Experienced a unilateral first stroke, either ischemic or hemorrhagic, in the carotid artery distribution.
* Diagnosed with stroke at least one month prior to participating in the study.
* Free from major post-stroke complications, such as recurrent stroke, hip fracture, or myocardial infarction.
* Residing within the community.
* Capable of ambulating 10 meters with or without the use of assistive devices.

Exclusion Criteria:

* Stroke secondary to subarachnoid hemorrhage or posterior circulation stroke.
* Life expectancy of less than one year.
* Comatose state.
* Inability to follow 3-step commands.
* Amputation.
* Poorly controlled diabetes, exemplified by conditions such as foot ulceration.
* Blindness.
* Progressive neurological diseases.
* Comprehensive aphasia.
* Medical instability.
* Significant musculoskeletal problems.
* Congestive cardiac failure.
* Unstable angina.
* Peripheral vascular disease.
* Neuropsychiatric disorders, including dementia, cognitive deficits, and severe depression.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with Kinematic representation of the temporal events during end-effector robot training | Pre-overground, Morning walk intervention, and post-overground of assessment in one day and will be recorded continuously for 20-30minutes
  The temporal events of foot position and foot pressure distributions will be identified from ground reaction forces (GRFs) during walking trials using the Tekscan In-shoes system (Tekscan, Inc., South Boston).
Muscle Activity in the lower extremities | Pre-overground, Morning walk intervention, and post-overground of assessment in one day and will be recorded continuously for 20-30minutes
  A wireless electromyographic sensor (Delsys Inc, Natick, MA) will be attached to the participant to analyze muscle activity in the lower extremities.
Spatiotemporal Patterns of Walking, Speeds | Pre-overground and post-overground of assessment in one day and will be recorded continuously for 20-30minutes
  Subjects will walk on an instrumented mat (Zeno Walkway) with the same model of New Balance shoes to measure self-selected and fastest comfortable speeds.
Spatiotemporal Patterns of Walking, Parameters | Pre-overground and post-overground of assessment in one day and will be recorded continuously for 20-30minutes
  Subjects will walk on an instrumented mat (Zeno Walkway) with the same model of New Balance shoes to measure the parameters during overground walking.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No